CLINICAL TRIAL: NCT00468936
Title: Open-Label, Randomized Study Comparing the Patient Reported Severity of GI Side Effects of MMF Versus EC-MPS in Maintenance Heart Transplant Patients.
Brief Title: Myfortic in Heart Transplant Patients With Gastrointestinal (GI) Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Dr Nadia Giannetti, McGill University Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMB 06-006; OCC 2006-104
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Heart Transplant Patients
Keywords: anti-rejection; GI side effects; heart transplant patients
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual medications (Cellcept)
- 2 (Active Comparator): Patients taking Myfortic
  Interventions: Drug: Myfortic

INTERVENTIONS:
Drug: Myfortic — enteric coated Cellcept pills in applicable dose for patient
  Arms: 2

SUMMARY:
Stable heart transplant patients on Mycophenolate Mofetil (MMF) will sign a screening consent form in order to be evaluated with the gastrointestinal symptom rating scale (GSRS) questionnaire. Those who score three or more on at least two questions are eligible for the study. Once they sign a study consent they are randomized to one of two arms. It is thought that the severity of GI side effects will be reduced over time in patients who are in the Myfortic arm versus the severity of GI side effects over time in patients who remain on MMF treatment. Patients are evaluated by GSRS, The Psychological Well-Being Schedule, and the IT01/02 Checklist for the evaluation of GI symptoms and followed for one year (visits 1 month, 3 months, 6 months, 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Stable dose MMF for at least 4 weeks
* Over 18 years of age
* Heart transplant at least three months prior to study

Exclusion Criteria:

* GI symptoms known not to be caused by MPA therapy
* Acute rejection episode in past 4 weeks
* History of malignancy since transplant
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
reduction in GSRS score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nadia S Giannetti, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada